CLINICAL TRIAL: NCT05923554
Title: Impact of Non-surgical Treatment of Peri-implant Mucositis on Incongruous Dental Prostheses Versus Congruous on a Single Tooth Restoration
Brief Title: Treatment of Peri-implant Mucositis on Incongruous Dental Prostheses Versus Congruous
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, Doctor, University of Catania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-150-PO
Record Dates: First submitted 2023-05-26; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Bleeding of Subgingival Space

STUDY DESIGN:
Intervention Model Description: After non-randomization, patients were assigned to a group with un-congruous single-tooth prostheses and a group with congruous single-tooth prostheses. Patients received a one-stage full-mouth scaling without chlorhexidine. Clinical and microbiological examination was performed at baseline, after 1, 2, and 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Un-congruous single tooth peri implantitis (Active Comparator): Patients were treated through non-surgical periodontal treatment for the peri-implant mucositis resolution
  Interventions: Other: Changes in Probing Depth to non-surgical periodontal therapy
- Congruous single tooth peri implantitis (Placebo Comparator): Patients were treated through non-surgical periodontal treatment for the peri implant mucositis resolution
  Interventions: Other: Changes in Probing Depth to non-surgical periodontal therapy

INTERVENTIONS:
Other: Changes in Probing Depth to non-surgical periodontal therapy — Changes in Probing Depth following non surgical periodontal treatment performed with hand and ultrasonic tips

SUMMARY:
The aim of the present study was to test the hypothesis that non-surgical periodontal therapy on peri-implant mucositis resolution results in a greater clinical improvement in patients with congruous versus non-congruous single dental implant restoration.

DETAILED DESCRIPTION:
The aim of the present study was to test the hypothesis that non-surgical periodontal therapy on peri-implant mucositis resolution results in a greater clinical improvement in patients with congruous versus non-congruous single dental implant restoration by comparing two groups of patients with peri-implant mucositis.

ELIGIBILITY:
Inclusion Criteria:

* peri-implant mucositis
* bleeding on probing and/or a gingival index <1 at least at one site at baseline
* absence of peri-implant bone loss during the last 2 years before baseline

Exclusion Criteria:

* Periodontal disease
* Systemic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing change % reduction | 6-months
  Reduction in bleeding on probing % change following non surgical periodontal therapy

SECONDARY OUTCOMES:
Reduction of probing depth in mm | 6-months
  Reduction of probing depth following non surgical periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Pubmed